CLINICAL TRIAL: NCT05865613
Title: Effect of Pulsed Electromagnetic Field Therapy on Headache, Fatigue, and CT Finding on Patients With Chronic Rhinosinusitis.
Brief Title: Effect of Electromagnetic Therapy on Patients With Chronic Rhinosinusitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: magnetic and rhinosinusitis
Record Dates: First submitted 2022-06-27; First posted 2023-05-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Magnetic Therapy; Rhinosinusitis; Headache; Fatigue
MeSH Terms: conditions — Rhinosinusitis; Headache; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic group (Experimental): Participants were randomized into either the PEMF group or sham treatment group by a computer-generated random number. The participants were treated using PEMF (20 G,7H for 10min). treatment was delivered for one month.
  Interventions: Device: Pulsed electromagnetic field
- Sham magnetic group (Sham Comparator): Participants were randomized into either the PEMF group or sham treatment group by a computer-generated random number. The participants were treated using PEMF without adjusting the output. treatment was delivered for one month.
  Interventions: Device: Pulsed electromagnetic field

INTERVENTIONS:
Device: Pulsed electromagnetic field — Participants were randomized into either the PEMF group or sham treatment group by a computer-generated random number. The participants were treated using PEMF (20 G ,7H for 10min) and sham treatment. treatment was delivered for one month.
  Other Names: Sham

SUMMARY:
This study aimed to evaluate the efficacy of Pulsed electromagnetic field (PEMF) for Chronic sinusitis in a randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Chronic sinusitis, or chronic rhinosinusitis, is an inflammatory condition defined by symptomatic inflammation of the paranasal sinuses lasting longer than 3 months. Common presenting symptoms include nasal obstruction, facial pressure or fullness, nasal discharge (anterior or posterior), and olfactory loss. Furthermore, chronic sinusitis is associated with reductions in patient quality of life, sleep quality, and daily productivity.

A pulsed electromagnetic field (PEMF) has an anti-inflammatory, antimicrobial, and improves the microcirculation of the mucosal membrane of the nasal cavity. It has been suggested that magnetic therapy can be used in treating chronic sinusitis but there is a scarce of studies about its usage.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from mild to moderate symptoms of rhinosinusitis.

Exclusion Criteria:

* pregnant or breastfeeding women.
* patients with definite deviated nasal septum, sinusitis, or history of operation within the last 6 months.
* patients with hypertension, diabetes mellitus, malignancy, active pulmonary tuberculosis, infection, active respiratory disease like asthma, or other systemic diseases.
* patients with long-term use of corticosteroids or immunosuppressive agents.
* patients who were involved in another clinical study within 30 days.
* patients who were unable to comply with the follow-up schedules.
* patients who had used antihistamines within 1 week, topical corticosteroids within 2 weeks, systemic corticosteroids within 4 weeks, anti-cholinergic drugs within 3 days, antileukotriene drugs within 1 week, decongestants within 3 days, tricyclic antidepressants or phenothiazines within 2 weeks, non-steroidal analgesics within 2 weeks, and other drugs which the researchers believed were inappropriate.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Headache | Baseline and one month.
  Headache was measured using VAS at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the headache.

SECONDARY OUTCOMES:
Fatigue | Baseline and one month.
  Fatigue was measured using fatigue scale at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the fatigue value
CT finding | Baseline and one month.
  Number of sinus opacifications before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo university, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No